CLINICAL TRIAL: NCT03448406
Title: A Phase III Randomised, Double-blind Trial to Evaluate the Effect of 12 Weeks Treatment of Once Daily EMPagliflozin 10 mg Compared With Placebo on ExeRcise Ability and Heart Failure Symptoms, In Patients With Chronic HeArt FaiLure With Preserved Ejection Fraction (HFpEF) (EMPERIAL - Preserved)
Brief Title: This Study Tests Empagliflozin in Patients With Chronic Heart Failure With Preserved Ejection Fraction (HFpEF). The Study Looks at How Far Patients Can Walk in 6 Minutes and at Their Heart Failure Symptoms.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1245-0167; 2017-004072-59 (EudraCT Number)
Record Dates: First submitted 2018-02-22; First posted 2018-02-28 (Actual); Results first posted 2020-12-08 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-11

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Empagliflozin (Experimental)
  Interventions: Drug: Empagliflozin
- Placebo (Active Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin — Film-coated tablet
  Other Names: JARDIANCE, JARDIANZ, GIBTULIO
  Arms: Empagliflozin
Drug: Placebo — Film-coated tablet
  Arms: Placebo

SUMMARY:
The primary objective of the study is to evaluate the effect of empagliflozin 10 mg versus placebo on exercise ability using the 6 minute walk test (6MWT) in patients with chronic heart failure (CHF) with preserved ejection fraction (LVEF > 40%).

Secondary objectives are to assess Patient-Reported Outcome (PRO)

ELIGIBILITY:
Inclusion Criteria:

* Of full age of consent (according to local legislation, usually ≥ 18 years) at screening.
* Male or female patients. Women of child bearing potential (WOCBP) must be ready and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria is provided in the patient information.
* Signed and dated written informed consent in accordance with ICHGCP and local legislation prior to admission to the trial
* Six minute walk test (6MWT) distance ≤350 m at screening and at baseline.
* Patients with CHF diagnosed for at least 3 months before Visit 1, and currently in NYHA class II-IV
* Chronic heart failure (CHF) with preserved Ejection fraction (EF) defined as left ventricle ejection fraction(LVEF) > 40 % as per echocardiography at Visit 1 per local reading and no prior measurement of LVEF ≤ 40% under stable conditions.
* Elevated N-Terminal Pro-Brain Natriuretic Peptide (NT-proBNP) > 300 pg/ml for patients without atrial fibrillation (AF), OR > 600 pg/ml for patients with AF, as analysed at the Central laboratory at Visit 1
* Patients must have at least one of the following evidence of heart failure (HF):

  * Structural heart disease (left atrial enlargement and/or left ventricular hypertrophy) documented by echocardiogram at Visit 1, OR
  * Documented Hospitalization for Heart Failure (HHF) within 12 months prior to Visit 1
* Consistent with prevailing CV guidelines, if oral diuretics are prescribed to control symptoms, patients must be on an appropriate and stable dose of oral diuretics for at least 2 weeks prior to Visit 1 to control symptoms.
* Clinically stable at randomization with no signs of heart failure decompensation (as per investigator judgement).

Exclusion Criteria:

* Myocardial infarction (increase in cardiac enzymes in combination with symptoms of ischaemia or newly developed ischaemic ECG changes), coronary artery bypass graft surgery or other major cardiovascular surgery, stroke or transient ischemic attack in past 90 days prior to Visit 1
* Acute decompensated HF (exacerbation of CHF) requiring intravenous (i.v.) diuretics, i.v. inotropes or i.v. vasodilators, or left ventricular assist device within 4 weeks prior to Visit 1, and/or during screening period until Visit 2
* Previous or current randomisation in another Empagliflozin Heart Failure trial (i.e. studies 1245.110, 1245.121, 1245-0168)
* Type 1 Diabetes Mellitus (T1DM)
* Impaired renal function, defined as eGFR < 20 mL/min/1.73 m2 (CKD-EPIcr) or requiring dialysis, as determined at Visit 1
* Symptomatic hypotension or a systolic blood pressure (SBP) < 100 mmHg at Visit 1 or 2
* SBP ≥ 180 mmHg at Visit 1 or 2, or SBP >160mmHg at both Visit 1 and 2
* Atrial fibrillation or atrial flutter with a resting heart rate > 110 bpm documented by ECG at Visit 1 (Screening)
* Unstable angina pectoris in past 30 days prior to Visit 1
* Largest distance walked in 6 minutes (6MWTD) at baseline <100m.
* Any presence of condition that precludes exercise testing such as:

  * claudication,
  * uncontrolled (according to investigator judgement) bradyarrhythmia or tachyarrhythmia,
  * significant musculoskeletal disease,
  * primary pulmonary hypertension,
  * severe obesity (body mass index ≥40.0 kg/m2),
  * orthopedic conditions that limit the ability to walk (such as arthritis in the leg, knee or hip injuries)
  * amputation with artificial limb without stable prosthesis function for the past 3 months
  * Any condition that in the opinion of the investigator would contraindicate the assessment of 6MWT
* Patients in a structured (according to Investigator judgement) exercise training program in the 1 month prior to screening or planned to start one during the course of this trial.
* ICD implantation within 1 month prior to Visit 1 or planned during the course of the trial
* Implanted cardiac resynchronisation therapy (CRT)
* Treatment with i.v. iron therapy or erythropoietin (EPO) within 3 months prior to screening.
* Further exclusion criteria applies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2019-10-04 (Actual); Study Completion 2019-10-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (108):
- United States (43):
  - Mobile Heart Specialists, PC, Mobile, Alabama
  - The Center for Clinical Trials, Inc., Saraland, Alabama
  - California Heart Specialists, Huntington Beach, California
  - Manshadi Heart Institute, Inc, Stockton, California
  - University of California Los Angeles, Torrance, California
  - University of Colorado Denver, Aurora, Colorado
  - Western Connecticut Health Network, Danbury, Connecticut
  - Infinite Clinical Research, Miami, Florida
  - Advance Medical Research Center, Miami, Florida
  - Bio1 Clinical Research, Miami Beach, Florida
  - Pharmacology Research, LLC, North Miami Beach, Florida
  - Palm Beach Gardens Research Center, LLC, Palm Beach Gardens, Florida
  - East Coast Institute for Research, LLC, Saint Augustine, Florida
  - Cozy Research LLC, Zephyrhills, Florida
  - Grady Memorial Hospital, Atlanta, Georgia
  - Georgia Arrhythmia Consultants and Research Institute, Warner Robins, Georgia
  - St Luke's Clinic - Idaho Cardiology Associates, Boise, Idaho
  - Northwest Heart Clinical Research, LLC, Arlington Heights, Illinois
  - Clinical Investigation Specialists, Inc, Gurnee, Illinois
  - Chicago Medical Research, Hazel Crest, Illinois
  - Midwest Heart and Vascular Specialists, Overland Park, Kansas
  - Grace Research, LLC, Bossier City, Louisiana
  - Grace Research, LLC, Shreveport, Louisiana
  - Clinical Trials of America LA, LLC, West Monroe, Louisiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - John D. Dingell VA Medical Center, Detroit, Michigan
  - Med Research One, Florissant, Missouri
  - Cox Medical Center South, Springfield, Missouri
  - The DOCS, Las Vegas, Nevada
  - Rutgers Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Albany Stratton VA Medical Center Albany, NY, Albany, New York
  - UNC REX Healthcare, Raleigh, North Carolina
  - PMG Research of Rocky Mount, LLC, Rocky Mount, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - Rama Research LLC, Marion, Ohio
  - Columbia Heart Clinic, Columbia, South Carolina
  - Black Hills Cardiovascular Research, Rapid City, South Dakota
  - The Jackson Clinic, PA, Jackson, Tennessee
  - DiscoveResearch, Inc., Beaumont, Texas
  - Angiocardiac Care of Texas, Houston, Texas
  - Acacia Medical Research Institute,LLC, Sugar Land, Texas
  - Mary Washington Hospital Research Department, Fredericksburg, Virginia
  - York Clinical Research, LLC, Norfolk, Virginia
- Australia (3):
  - Canberra Hospital, Garran, Australian Capital Territory
  - University of the Sunshine Coast, Birtinya, Queensland
  - Peninsular Health CV Research Unit, Frankston, Victoria
- Canada (4):
  - University of Calgary, Calgary, Alberta
  - KMH Cardiology Centres Inc., Mississauga, Ontario
  - Toronto Heart Centre, Toronto, Ontario
  - Sameh Fikry Medicine Professional Corporation, Waterloo, Ontario
- Germany (13):
  - CIMS Studienzentrum Bamberg GmbH, Bamberg
  - Klinische Forschung Berlin GbR, Berlin
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Köln (AöR), Cologne
  - Cardiologicum Dresden und Pirna, Dresden
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - IKF Pneumologie GmbH & Co. KG, Frankfurt
  - Universitäts-Herzzentrum Freiburg, Bad Krozingen GmbH, Freiburg im Breisgau
  - Universitätsklinikum Leipzig, Leipzig
  - Universitätsklinikum Magdeburg AöR, Magdeburg
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Universitätsklinikum Ulm, Ulm
  - Universitätsklinikum Würzburg, Würzburg
- Greece (6):
  - General Hospital of Athens Konstantopoulio-Agia Olga, Athens
  - General Hospital of Athens "G. Gennimatas", Athens
  - General Hospital of Chalkida, Chalcis
  - University General Hospital of Heraklion, Herakleion, Crete
  - Univ. Gen. Hosp. of Ioannina, Ioannina
  - University Hospital of Thessaloniki AHEPA, Thessaloniki
- Italy (7):
  - Centro Cardiologico Monzino-IRCCS, Milan
  - Asst Santi Paolo E Carlo, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Ospedale Regina Montis Regalis, Mondovì (CN)
  - Università Federico II, Napoli
  - Università degli studi di Palermo, Palermo
  - IRCCS San Raffaele, Roma
- Norway (4):
  - Sykehuset Østfold Kalnes, Grålum
  - Oslo Universitetssykehus HF, Rikshospitalet, Oslo
  - Helse Stavanger, Stavanger Universitetssykehus, Stavanger
  - St. Olavs Hospital, Universitetssykehuset i Trondheim, Trondheim
- Poland (9):
  - INTERCORE Medical Center, Bydgoszcz
  - 10.Military Clin.Hospital&Polyclinic, Bydgoszcz
  - Leszek Bryniarski Specialized Medical Cabinet, Krakow
  - Card.Cli.Mil.Med.Ac.Uni.Cli.Hosp. Cent.Vetera.Hosp.Lodz, Lodz
  - Cent.Clin.Hosp.Med.Univ.Lodz,Electrocard, Lodz
  - Provincial Specialist M. Kopernik Hospital, Lodz
  - Independent Public Healthcare, Dept. of Cardiology, Pulawy, Puławy
  - Central Hospital of Medical Academy, Warsaw, Warsaw
  - 4. Military Clinical Hospital with Polyclinic SP ZOZ, Wroclaw
- Portugal (7):
  - CHLO, EPE - Hospital de Santa Cruz, Carnaxide
  - CHUC - Centro Hospitalar e Universitário de Coimbra, EPE, Coimbra
  - Centro Hosp. de Leiria-Pombal, Leiria
  - CHLC, EPE - Hospital de Santa Marta, Lisbon
  - CHLO, EPE - Hospital S. Francisco Xavier, Lisbon
  - CHULN, EPE - Hospital de Santa Maria, Lisbon
  - Centro Hospitalar Universitário São João,EPE, Porto
- Spain (8):
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital San Rafael, Granada
  - Hospital de la Inmaculada Concepción, Granada
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital La Princesa, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Clínico de Valencia, Valencia
- Sweden (4):
  - Sahlgrenska US, Göteborg, Gothenburg
  - Sahlgrenska Universitetssjukhuset, Östra, Gothenburg
  - Skånes universitetssjukhus, Lund, Lund
  - Akardo Med Site, Stockholm

REFERENCES:
- [Derived] Anker SD, Ponikowski P, Wanner C, Pfarr E, Hauske S, Peil B, Salsali A, Ritter I, Koitka-Weber A, Brueckmann M, Lindenfeld J, Abraham WT; EMPERIAL Investigators and National Coordinators. Kidney Function After Initiation and Discontinuation of Empagliflozin in Patients With Heart Failure With and Without Type 2 Diabetes: Insights From the EMPERIAL Trials. Circulation. 2021 Oct 12;144(15):1265-1267. doi: 10.1161/CIRCULATIONAHA.121.054669. Epub 2021 Aug 16. No abstract available. PMID 34397263
- [Derived] Abraham WT, Ponikowski P, Brueckmann M, Zeller C, Macesic H, Peil B, Brun M, Ustyugova A, Jamal W, Salsali A, Lindenfeld J, Anker SD; EMPERIAL Investigators and National Coordinators. Rationale and design of the EMPERIAL-Preserved and EMPERIAL-Reduced trials of empagliflozin in patients with chronic heart failure. Eur J Heart Fail. 2019 Jul;21(7):932-942. doi: 10.1002/ejhf.1486. Epub 2019 Jun 19. PMID 31218819
- [Derived] Nassif ME, Kosiborod M. Effects of sodium glucose cotransporter type 2 inhibitors on heart failure. Diabetes Obes Metab. 2019 Apr;21 Suppl 2:19-23. doi: 10.1111/dom.13678. PMID 31081589

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Randomised, double-blind, placebo-controlled, parallel-group trial in patients with chronic Heart Failure with preserved Ejection Fraction (HFpEF) to evaluate the effect of Empagliflozin versus Placebo on exercise and heart failure symptoms.
Pre-assignment Details: Only subjects that met all the study inclusion and none of the exclusion criteria were to be entered in the study. All subjects were free to withdraw from the clinical trial at any time for any reason given. Close monitoring of all subjects was adhered to throughout the trial conduct.
Groups:
- Placebo: 1 film-coated tablet of Placebo matching Empagliflozin was administered orally once daily for 12 weeks in participants with chronic Heart Failure (CHF) with preserved ejection fraction (LVEF > 40%).
- 10 mg Empagliflozin: 1 film-coated tablet of 10 milligram (mg) of Empagliflozin was administered orally once daily for 12 weeks in participants with chronic Heart Failure (CHF) with with preserved ejection fraction (LVEF > 40%).
Period: Overall Study
Arm/Group | Placebo | 10 mg Empagliflozin
Started | 158 | 157
Completed | 147 | 144
Not Completed | 11 | 13
Not completed — Noncompliance of scheduled visits | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Adverse Event | 8 | 9

BASELINE CHARACTERISTICS:
Population: Randomised Set: All randomised participants, regardless of whether treated or not.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 10 mg Empagliflozin | Total
Number analyzed (Participants) | 158 | 157 | 315
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.9 (8.6) | 73.0 (9.0) | 73.5 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 70 | 136
  Male | 92 | 87 | 179
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 18 | 37
  Not Hispanic or Latino | 139 | 138 | 277
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 13 | 32
  White | 135 | 140 | 275
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 1 | 1
Exercise capacity as measured by the 6-Minutes-Walking-Test (6MWT) distance at baseline [Median (Inter-Quartile Range); unit: Meter] — 6 Minute Walking test measures the distance walked in 6 minutes in standardised conditions at baseline.
  Meter | 299.5 [245.0 to 331.0] | 297.0 [246.0 to 326.0] | 299.0 [245.0 to 330.0]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in Exercise Capacity as Measured by the Distance Walked in 6 Minutes in Standardised Conditions (6MWTD)
Description: Change from baseline to week 12 in exercise capacity as measured by the distance walked in 6 minutes in standardised conditions (6MWTD). If repeated 6-minutes walk test (6MWT) measurements were available for the same day, the longest distance was used for analysis. Change from baseline was defined as the distance walked in 6 minutes at Week 12 minus the baseline value.
  Baseline value was defined as the last available measurement before start of treatment with randomised study medication. If a participant was present at the visit at Week 12 but did not perform the 6MWT, the participant was evaluated as having walked a distance of 0 meter. If no value was available for Week 12, an imputed value was used. Patients with missing week 12 data who had no clinical event were ranked below any patient with non-missing data, but above the patients who had clinical events. Patients who died before week 12 were ranked below the patients in all categories above.
Time Frame: At baseline and at Week 12
Population: Randomised Set: All participants that were randomised, regardless of whether treated or not.
Measure: Median (Inter-Quartile Range); unit: Meter (m)
Arm/Group | Placebo | 10 mg Empagliflozin
Number analyzed (Participants) | 158 | 157
Meter (m) | 5.0 [-20.0 to 33.0] | 10.0 [-10.0 to 32.0]
Statistical Analysis 1: Comparison: Placebo vs 10 mg Empagliflozin; H0: There is no difference between the effect of Placebo and the effect of empagliflozin; Test type: Superiority; p = 0.3660, Wilcoxon rank test, normal approximation; Median difference (HL-estimate) = 4.0, 95% CI 2-sided [-5.0 to 13.0] — Empagliflozin vs. Placebo. For estimation of effect, the non-parametric Hodge-Lehman (HL) estimate for the median difference was calculated

2. Secondary Outcome: Change From Baseline to Week 12 in Kansas City Cardiomyopathy Questionnaire (KCCQ) Total Symptom Score (TSS)
Description: Change from baseline in KCCQ-TSS was defined as the endpoint value at week 12 minus the last available measurement before start of treatment with randomised study medication. The KCCQ is 23 item self-administered questionnaire and comprises 7 domains: physical limitation, symptom frequency, symptom burden, symptom stability, social limitation, self-efficacy and quality of life. Additionally 3 summary scores exist: TSS, clinical summary score, and overall summary score. The scores of the KCCQ domains and summary scores range from 0 to 100, with higher score indicating better outcome. If no questionnaire was available at week 12, an imputed value was used. Patients with missing week 12 data who had no clinical event were ranked below any patient with non-missing data, but above the patients who had clinical events. Patients who died before week 12 were ranked below the patients in all categories above. If no questionnaire was available at baseline, change from baseline was not imputed.
Time Frame: At baseline and at Week 12
Population: Randomised Set: All participants that were randomised, regardless of whether treated or not.
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | Placebo | 10 mg Empagliflozin
Number analyzed (Participants) | 158 | 157
Score on a scale | 2.08 [-6.25 to 20.83] | 4.17 [-3.13 to 16.67]
Statistical Analysis 1: Comparison: Placebo vs 10 mg Empagliflozin; H0: There is no difference between the effect of Placebo and the effect of empagliflozin; Test type: Superiority; p = 0.2783, Wilcoxon rank test, normal approximation; Median difference (HL-estimate) = 2.08, 95% CI 2-sided [-2.08 to 6.25] — Empagliflozin vs. Placebo. For estimation of effect, the non-parametric Hodges-Lehmann estimate for the median difference was calculated

3. Secondary Outcome: Change From Baseline to Week 12 in Chronic Heart Failure Questionnaire Self- Administered Standardized Format (CHQ-SAS) Dyspnea Score
Description: Change from baseline in CHQ-SAS was defined as the endpoint value at week 12 minus the last available endpoint value before start of treatment with randomised study medication. The CHQ-SAS evaluates 3 domains: dyspnoea, fatigue, and emotional function. Scores of the domains range from 1 to 7, with higher score indicating better quality of life. If no questionnaire was available at week 12, an imputed value was used. Patients with missing week 12 data who had no clinical event were ranked below any patient with non-missing data, but above the patients who had clinical events. Patients who died before week 12 were ranked below the patients in all categories above. If no questionnaire was available at baseline, change from baseline was not imputed.
Time Frame: At baseline and at Week 12
Population: Participants in the randomised set (RS) who have no missing values at baseline.
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | Placebo | 10 mg Empagliflozin
Number analyzed (Participants) | 158 | 156
Score on a scale | 0.20 [-0.40 to 1.00] | 0.10 [-0.40 to 1.00]
Statistical Analysis 1: Comparison: Placebo vs 10 mg Empagliflozin; H0: There is no difference between the effect of Placebo and the effect of empagliflozin; Test type: Superiority; p = 0.5512, Wilcoxon rank test, normal approximation; Median difference (HL-estimate) = -0.07, 95% CI 2-sided [-0.35 to 0.20] — Empagliflozin vs. Placebo. For estimation of effect, the non-parametric Hodges-Lehmann (HL) estimate for the median difference was calculated

4. Secondary Outcome: Change From Baseline to Week 6 in Exercise Capacity as Measured by the Distance Walked in 6 Minutes
Description: Change from baseline to week 6 in exercise capacity as measured by the distance walked in 6 minutes in standardised conditions. Change from baseline was defined as the distance walked in 6 minutes at Week 6 minus the baseline value. Baseline value was defined as the last available measurement before start of treatment with randomised study medication.
  If a participant was present at the visit at Week 6 but did not perform the 6-Minuted Walking Test, the participant was evaluated as having walked a distance of 0 meter. If no value was available for Week 6, an imputed value was used.
Time Frame: At baseline and at Week 6
Population: Randomised Set: All participants that were randomised, regardless of whether treated or not.
Measure: Median (Inter-Quartile Range); unit: Meter (m)
Arm/Group | Placebo | 10 mg Empagliflozin
Number analyzed (Participants) | 158 | 157
Meter (m) | 1.0 [-17.0 to 21.0] | 7.0 [-14.0 to 23.0]
Statistical Analysis 1: Comparison: Placebo vs 10 mg Empagliflozin; H0: There is no difference between the effect of Placebo and the effect of empagliflozin; Test type: Superiority; p = 0.3657, Wilcoxon rank test, normal approximation; Median Difference (HL-estimate) = 3.0, 95% CI 2-sided [-4.0 to 11.0] — [estimate comment as in outcome 3, analysis 1]

5. Secondary Outcome: Change From Baseline in Clinical Congestion Score at Week 12
Description: Change from baseline to week 12 in Clinical Congestion score is defined as the score-value at week 12 minus the score-value at baseline. Baseline value was defined as the last available measurement before start of treatment with randomised study medication. The Clinical Congestion Score (summary score) is based on 3 items: orthopnoea, jugular venous distention (JVD) and oedema. Each item was assessed through a 4-measure questionnaire, which was further converted to a standardised 4-point scale ranging from 0 to 3, with 0 indicating no or fewer symptoms and 3 indicating continous or more symptoms. If at least 2 of the 3 items are not missing, the summary score is calculated as: (average over items JVD, orthopnea and oedema actually answered)*3. The summary score ranges from 0 to 9, with lower value indicating better health, and higher value indicating worse health. Mean is adjusted mean.
Time Frame: At baseline and at Week 12
Population: Only participants in the randomised set (RS) who have values at baseline and at week 12.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Placebo | 10 mg Empagliflozin
Number analyzed (Participants) | 155 | 156
Score on scale | -0.28 (0.08) | -0.36 (0.08)
Statistical Analysis 1: Comparison: Placebo vs 10 mg Empagliflozin; Test type: Other; p = 0.4440, Mixed Model Repeated Measure (MMRM); Covariates: visit-by-treatment interaction, baseline-by-visit interaction. Unstructured covariance structure was used to model within-patient errors; Difference of adjusted mean = -0.09, 95% CI 2-sided [-0.31 to 0.14], Standard Deviation 0.11

6. Secondary Outcome: Change From Baseline in Patient Global Impression of Severity (PGI-S) of Heart Failure Symptoms at Week 12
Description: Change from baseline to week 12 in PGI-S of Heart Failure Symptoms. The Patient Global Impression of Severity (PGI-S) of Heart Failure Symptoms is a 1-item questionnaire to assess the patient's impression of symptoms severity, specifically: shortness of breath, fatigue and swelling. The PGI-S asks the Patient to choose one response that best describes how his/her heart failure symptoms, specifically: shortness of breath, fatigue and swelling are now on a 5-category scale, ranging from 'Not at all' (1) to 'Very severe' (5). Number of participants by change in score are reported. Change in score was defined as the number of categories improved/deteriorated from baseline to week 12.
Time Frame: At baseline and at Week 12
Population: Only participants in the randomised set (RS) who have values at baseline and at week 12.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 10 mg Empagliflozin
Number analyzed (Participants) | 154 | 153
Participants
  4 categories improvement | 1 | 0
  3 categories improvement | 2 | 1
  2 categories improvement | 11 | 8
  1 category improvement | 46 | 42
  No change | 70 | 79
  1 category deterioration | 17 | 16
  2 categories deterioration | 6 | 6
  3 categories deterioration | 0 | 1
  4 categories deterioration | 1 | 0
Statistical Analysis 1: Comparison: Placebo vs 10 mg Empagliflozin; Test type: Other; p = 0.3924, Cochran-Mantel-Haenszel test; Test on difference in mean treatment scores, based on modified ridit scores

7. Secondary Outcome: Change From Baseline in Patient Global Impression of Severity (PGI-S) of Dyspnea Severity at Week 12
Description: Change from baseline to week 12 in Patient Global Impression of Severity (PGI-S) of dyspnoea. The PGI-S of Dyspnoea is a 1-item questionnaire designed to assess the participant´s impression of symptom severity, specifically dyspnoea. The PGI-S item asks the participant to choose one response that best describes how his/her dyspnoea is now on a 5-category scale, ranging from 'Not at all' (1) to 'Very severe' (5). Number of participants by change in score are reported. Change in score was defined as the number of categories improved/deteriorated from baseline to week 12.
Time Frame: At baseline and at Week 12
Population: Only participants in the randomised set (RS) who have values at baseline and at week 12.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 10 mg Empagliflozin
Number analyzed (Participants) | 154 | 153
Participants
  4 categories improvement | 1 | 0
  3 categories improvement | 4 | 1
  2 categories improvement | 8 | 13
  1 category improvement | 45 | 48
  No change | 70 | 70
  1 category deterioration | 18 | 20
  2 categories deterioration | 7 | 1
  3 categories deterioration | 1 | 0
  4 categories deterioration | 0 | 0
Statistical Analysis 1: Comparison: Placebo vs 10 mg Empagliflozin; Test type: Other; p = 0.4435, Cochran-Mantel-Haenszel test; Test on difference in mean treatment scores, based on modified ridit scores

8. Secondary Outcome: Patient Global Impression of Change (PGI-C) in Heart Failure Symptoms at Week 12
Description: The Patient Global Impression of Change (PGI-C) in Heart Failure Symptoms is a 1-item questionnaire to assess the patient's impression of change in heart failure symptoms, specifically: shortness of breath, fatigue, and swelling. The PGI-C asks the patient to choose one Response that best describes the overall change (if any) in his/her heart failure symptoms, specifically: shortness of breath, fatigue, and swelling since he/she started taking the study medication on a 7- category scale ranging from 'Very much better' (+3) to 'Very much worse' (-3).
Time Frame: Week 12
Population: Only participants in the randomised set (RS) who have values at week 12.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 10 mg Empagliflozin
Number analyzed (Participants) | 154 | 153
Participants
  Very much worse | 1 | 0
  Much worse | 0 | 3
  A little worse | 11 | 7
  No change | 62 | 55
  A little better | 41 | 48
  Much better | 31 | 35
  Very much better | 8 | 5
Statistical Analysis 1: Comparison: Placebo vs 10 mg Empagliflozin; Test type: Other; p = 0.5124, Cochran-Mantel-Haenszel test; Test on difference in mean treatment scores, based on modified ridit scores

9. Secondary Outcome: Patient Global Impression of Change (PGI-C) in Dyspnea at Week 12
Description: The PGI-C in Dyspnoea is a 1-item questionnaire designed to assess the patient's Impression of change in dyspnoea. The PGI-C asks the patient to choose one response that best describes the change (if any) in his/her shortness of breath when performing usual activities since he/she started taking the study medication on a 7-category scale ranging from 'Very much better' (+3) to 'Very much worse' (-3).
Time Frame: Week 12
Population: Only participants in the randomised set (RS) who have values at week 12.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 10 mg Empagliflozin
Number analyzed (Participants) | 154 | 153
Participants
  Very much worse | 0 | 0
  Much worse | 2 | 3
  A little worse | 6 | 7
  No change | 72 | 57
  A little better | 32 | 45
  Much better | 31 | 36
  Very much better | 11 | 5
Statistical Analysis 1: Comparison: Placebo vs 10 mg Empagliflozin; Test type: Other; p = 0.5713, Cochran-Mantel-Haenszel test; Test on difference in mean treatment scores, based on modified ridit scores

10. Secondary Outcome: Relative Change From Baseline in N-terminal Pro-brain Natriuretic Peptide (NTproBNP) at Week 12
Description: Relative change from baseline to week 12 in N-terminal pro-brain natriuretic peptide (NTproBNP). Relative change from baseline is expressed as ratio of week 12 to baseline. Baseline value was defined as the mean of all available measurements from the screening visit until start of treatment with randomised study medication. Mean is adjusted mean.
Time Frame: Within 3 weeks prior to treatment start and at Week 12.
Population: Only participants in the randomised set (RS) who had values at baseline and at week 12.
Measure: Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Placebo | 10 mg Empagliflozin
Number analyzed (Participants) | 155 | 156
Ratio | 1.04 [0.96 to 1.13] | 0.99 [0.92 to 1.08]
Statistical Analysis 1: Comparison: Placebo vs 10 mg Empagliflozin; Test type: Other; p = 0.4032, Mixed model repeated Measure (MMRM); Covariates: Visit-by-treatment interaction and baseline-by-visit interaction. Unstructured covariance structure to model within-patient errors; Adjusted geometric mean ratio = 0.95, 95% CI 2-sided [0.85 to 1.07] — Adjusted geometric mean ratio [Empagliflozin/Placebo] of relative change to baseline

ADVERSE EVENTS:
Time Frame: From first intake of study medication, until 7 days after last intake of study medication, up to 92 days.
Description: Treated Set: All participants who were treated with at least one dose of study medication.
Arm/Group | Placebo | 10 mg Empagliflozin
All-Cause Mortality (participants affected / at risk) | 0/158 | 1/157
Serious Adverse Events (participants affected / at risk) | 29/158 | 20/157
Other Adverse Events (participants affected / at risk) | 0/158 | 0/157
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=158) | 10 mg Empagliflozin (N=157)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 2
Atrial flutter (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 13 | 6
Pericarditis (Cardiac disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Generalised oedema (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1
Hepatic haemorrhage (Hepatobiliary disorders) | 1 | 0
Hepatic mass (Hepatobiliary disorders) | 1 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0
Asymptomatic bacteriuria (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Helicobacter duodenitis (Infections and infestations) | 0 | 1
Helicobacter gastritis (Infections and infestations) | 0 | 1
Necrotising fasciitis (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Blood glucose increased (Investigations) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain injury (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Anuria (Renal and urinary disorders) | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 0
Haemorrhage urinary tract (Renal and urinary disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-10-21): https://cdn.clinicaltrials.gov/large-docs/06/NCT03448406/SAP_000.pdf
  • Study Protocol (2018-05-16): https://cdn.clinicaltrials.gov/large-docs/06/NCT03448406/Prot_001.pdf